CLINICAL TRIAL: NCT03590691
Title: Conquering Hypertension in Vietnam: Solutions at Grassroots Level
Acronym: HY-TREC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Vietnam (Other Government)
Collaborators: University of Massachusetts, Worcester (Other); Baylor Research Institute (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Tran Thi Mai Oanh, Principal Investigator, Director of Health Strategy and Policy Institute, Ministry of Health, Vietnam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 5552338110000; 1U01HL138631-01 (NIH)
Record Dates: First submitted 2018-05-31; First posted 2018-07-18 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Hypertension
Keywords: storytelling
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: A cluster-randomized trial design
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison group (Active Comparator): Vietnam National Hypertension Program: a training program for health care workers and a health educational program for general public.
  Interventions: Other: Vietnam National Hypertension Program
- Intervention group (Experimental): Vietnam National Hypertension Program including training program for health care workers and an health educational program for general public.
  PLUS
  Three selected enhancements integrated into routine clinical care:
  1. expanded community health worker services;
  2. home blood pressure self-monitoring; and
  3. a "storytelling intervention".
  Interventions: Other: Vietnam National Hypertension Program; Other: Expanded community health worker services; Behavioral: Storytelling intervention; Behavioral: Home blood pressure self-monitoring

INTERVENTIONS:
Other: Vietnam National Hypertension Program — A training program for health care workers including physicians and nurses and a health educational program for general public regarding hypertension management at community level will be implemented
Other: Expanded community health worker services — A training program will be implemented for community health workers regarding hypertension management at community level so that they can assist patients better manage their blood pressure at home.
  Arms: Intervention group
Behavioral: Storytelling intervention — The storytelling intervention consists of interactive, literacy-appropriate, and culturally sensitive multimedia storytelling modules for motivating behavior change through the power of patients speaking in their own voice. Based on preferences that emerged during the researchers' formative work with the partnering rural communities, the storytelling intervention will be delivered by DVD, with serial installments at baseline and at 3, 6, and 12 months after trial enrollment.
  Arms: Intervention group
Behavioral: Home blood pressure self-monitoring — Patients with hypertension will be provided blood pressure monitors and guided to self-measure their blood pressure and to record their blood pressure daily at home.
  Arms: Intervention group

SUMMARY:
The objectives of the proposed project are to evaluate the implementation and effectiveness of two multi-faceted community and clinic-based strategies on the control of elevated blood pressure (BP) among adults in Vietnam via a cluster-randomized trial design.

Sixteen communities will be randomized to either an intervention (8 communities) or comparison group (8 communities). Eligible and consenting adult study participants with HTN (n = 680) will be assigned to intervention/comparison status based on the community in which they reside.

DETAILED DESCRIPTION:
"Đương đầu với bệnh Tăng huyết áp ở Việt Nam: Giải pháp từ Y tế cơ sở (Conquering Hypertension in Vietnam: Solutions at Grassroots level)" (Vietnam Hy-TREC) Background: Similar to other low- and middle-income countries, Vietnam has been experiencing an epidemiologic transition with an increasing burden of non-communicable diseases (NCD). The key risk factors for cardiovascular disease (CVD) are either on the rise or at alarming levels in Vietnam, particularly hypertension (HTN). Inasmuch, the burden of CVD will continue to increase in Vietnamese men and women unless effective prevention and control measures are put in place.

Objectives: This project will be evaluating the implementation and effectiveness of two multi-faceted community and clinic-based strategies for the control of hypertension among adults residing in the rural Red River Delta region of Vietnam with uncontrolled hypertension through use of a cluster-randomized trial design.

Study population:Sixteen communities will be randomized to either an intervention (8 communities) or comparison group (8 communities). Eligible and consentingadult study participants with uncontrolled HTN (n = 680) will be assigned to intervention/comparison status based on the community in which they reside.

Methods: Both comparison and intervention groups will receive a multi-level intervention modeled after the Vietnam National Hypertension Program. Components of this program include education and practice change modules for health care providers, accessible reading materials for patients, and a community awareness multi-media program. In addition to the Vietnam National Hypertension Program, the intervention group only will receive three carefully selected enhancements integrated into routine clinical care: (1) expanded community health worker services; (2) home blood pressure self-monitoring; and (3) a "storytelling intervention," previously developed and pilot tested for feasibility and effectiveness by members of the research team. The storytelling intervention consists of interactive, literacy-appropriate, and culturally sensitive multimedia storytelling modules for motivating behavior change through the power of patients speaking in their own voice. Based on preferences that emerged during our formative work with our partnering rural communities, the storytelling intervention will be delivered by DVD, with serial installments at baseline and again at 3, 6, and 12 months after trial enrollment. Differences in changes in blood pressure and other factors will be assessed in both study groups at several follow-up time points. In conjunction with the work done being accomplished during the pilot feasibility study, current efforts by the Vietnam National Hypertension Program, and the proposed investigation, this project addresses a serious clinical and public health problem in Vietnam by implementing the first community-based study using a culturally-literacy appropriate intervention to control elevated blood pressure among the adult Vietnamese population.

ELIGIBILITY:
Inclusion Criteria:

1. residence in a study commune;
2. at least 25 years old;
3. presence of uncontrolled HTN based on the screening process described previously and
4. willingness to provide informed consent.

Exclusion Criteria:

1. participation in another hypertension research study;
2. pregnant;
3. advanced cognitive impairment; or
4. previous participation in developing or having exposure to the hypertension storytelling modules.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 671 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in systolic blood pressure at 12 months | At baseline and at 3, 6, and 12 months after trial enrollment
  Changes in systolic blood pressure will be assessed in both study groups at several follow-up time points.

SECONDARY OUTCOMES:
Change from baseline in diastolic blood pressure at 12 months | At baseline and at 3, 6, and 12 months after trial enrollment
  Changes in diastolic blood pressure will be assessed in both study groups at several follow-up time points.
Change from baseline in medication adherence self-efficacy score at 12 months | At baseline and 12 months after trial enrollment
  Patients medication adherence self-efficacy will be measured using the Medication Adherence Self-efficacy Scale (MASES) instrument.
Changes from the baseline in proportions of patients with risk factors for CVD at 12 months | At baseline and 12 months after trial enrollment
  WHO STEPs questionnaires will be used to collect data on risk factors for CVD including tobacco use, alcohol consumption, salt intake and physical activities. Proportions of patients with current smoking, excessive use of alcohol, high salt intake, and low physical activity will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Tran Thi Mai Oanh, PhD, Principal Investigator — Health Strategy and Policy Institute
Locations (1):
- Health Strategy and Policy Institute, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen HL, Ha DA, Tran OT, Phan VH, Nguyen CT, Nguyen GH, Nguyen TT, Le TT, Goldberg RJ, Wang B, Tang ET, Chiriboga G, Budhwani H, Allison JJ. Conquering hypertension in Vietnam: 12- month follow up results from a cluster-randomised controlled trial. Lancet Reg Health West Pac. 2024 Jul 1;48:101123. doi: 10.1016/j.lanwpc.2024.101123. eCollection 2024 Jul. PMID 39045484
- [Derived] Nguyen HL, Tran OT, Ha DA, Phan VH, Nguyen CT, Nguyen GH, Nguyen TT, Chiriboga G, Goldberg RJ, Allison JJ. Impact of the COVID-19 pandemic on clinical research activities: Survey of study participants and health care workers participating in a hypertension trial in Vietnam. PLoS One. 2021 Jul 15;16(7):e0253664. doi: 10.1371/journal.pone.0253664. eCollection 2021. PMID 34264973
- [Derived] Ha DA, Tran OT, Nguyen HL, Chiriboga G, Goldberg RJ, Phan VH, Nguyen CT, Nguyen GH, Pham HV, Nguyen TT, Le TT, Allison JJ. Conquering hypertension in Vietnam-solutions at grassroots level: study protocol of a cluster randomized controlled trial. Trials. 2020 Nov 27;21(1):985. doi: 10.1186/s13063-020-04917-8. PMID 33246495